CLINICAL TRIAL: NCT07147920
Title: Clinical Validation of the Perin Health Patch Electrocardiogram Monitoring Device: A Multi-Component Study Evaluating Signal Quality, Placement Tolerance, and Long-Term Performance
Brief Title: Validation of Perin Health Patch ECG Monitoring Device Performance and Placement Accuracy
Status: Completed | Type: Observational
Sponsor: Perin Health Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-25-001
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: ECG; Electrocardiography; Monitoring, Physiologic
Keywords: ECG validation study; electrocardiogram accuracy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Chest-Worn ECG Monitoring Device — The Perin Health Patch is a non-invasive, chest-worn wearable device designed to continuously monitor electrocardiogram (ECG) signals using dry conductive adhesive electrodes. In this validation study, the device will be evaluated for its ability to accurately measure ECG parameters including heart rate, QT interval, QRS duration, and R-R intervals compared to FDA-cleared Holter monitors.
  The study intervention involves three components: (1) simultaneous ECG recording with the patch and reference Holter monitor for 15 minutes while participants remain seated, (2) placement tolerance testing where the patch is positioned at various locations (±20mm from optimal placement) to assess performance under suboptimal positioning, and (3) long-term wear evaluation where participants wear the patch continuously for 15 days with periodic assessments. The intervention is limited to device application and ECG data collection under controlled conditions, with no therapeutic treatment provided.

SUMMARY:
The goal of this clinical trial is to test how accurately and reliably a new chest-worn device called the Perin Health Patch measures heart rhythms (ECG) in adults aged 22 and older. The main questions it aims to answer are:

* How accurately does the Perin Health Patch measure heart rhythm compared to standard hospital ECG monitoring equipment?
* Does the patch still work properly if it's placed slightly off from the exact recommended position on the chest?
* Does the patch maintain good performance when worn continuously for 15 days?

The study has three parts that test different aspects of the device. Participants will:

* Wear the Perin Health Patch on their chest along with standard ECG monitoring equipment for comparison
* Have ECG recordings taken while sitting quietly for 15 minutes
* For the placement study: have the patch placed in several different positions to test if small placement errors affect performance
* For the long-term study: wear the patch continuously for 15 days at home with regular check-ups on days 1, 7, 10, and 15

The study will include both healthy adults and people with heart or lung conditions like heart failure, COPD, high blood pressure, or diabetes to test how well the device works for different types of patients. Researchers will compare the heart rhythm measurements from the chest patch to standard medical monitoring equipment to determine if the patch is accurate enough for medical use. Some participants will complete just one part of the study, while others may participate in multiple parts depending on which aspect of the device is being tested.

ELIGIBILITY:
Inclusion Criteria:

* Adults 22 to 90 years of age
* Healthy or chronic cardiopulmonary conditions or recent procedures
* Able to comply with study procedure

Exclusion Criteria:

* Pediatric or adolescent patients (age ≤21 years)
* Pacemaker
* A history of skin reactions to medical adhesives
* Any psychosocial condition or circumstance that, in the opinion of the investigator, would interfere with the conduct of the study or the patient's care and/or safety
* Pregnant
* Current participation in any other clinical study
* Refusal to participate

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from multiple clinical sites including hospital settings, clinical research facilities, and home healthcare providers. The population includes both healthy adult volunteers and patients with chronic cardiovascular or pulmonary conditions such as COPD, congestive heart failure, hypertension, coronary artery disease, chronic kidney disease, and diabetes. Recruitment targets a demographically diverse sample representative of the intended use population for remote cardiac monitoring, with specific attention to age, sex, BMI, and racial/ethnic diversity to ensure robust validation across patient subgroups commonly encountered in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
ECG Timing Interval Equivalence Between Perin Health Patch and Reference Holter Monitor | During single 15-minute recording session and up to 15 days of continuous monitoring
  Equivalence of ECG measurements between the investigational chest patch and FDA-cleared Holter monitor using Two One-Sided Tests (TOST) statistical methodology. ECG recordings are taken simultaneously from both devices while participants sit quietly for comparison. Equivalence is demonstrated when confidence intervals for mean differences fall within pre-specified clinical margins for key ECG timing intervals including QT interval, QRS duration, and R-R interval. Signal morphology similarity is assessed using Pearson correlation coefficient (where 1.0 indicates perfect similarity) and normalized root mean square error (where 0% indicates identical signals).

SECONDARY OUTCOMES:
Heart Rate Measurement Accuracy | During single 15-minute recording session and up to 15 days of continuous monitoring
  Accuracy of heart rate measurements from the investigational device compared to the reference Holter monitor. Heart rate is calculated from R-R intervals during simultaneous ECG recordings. Accuracy is assessed using mean absolute error between devices, where lower values indicate better agreement.
ECG Signal Quality Equivalence | During single 15-minute recording session and up to 15 days of continuous monitoring
  Comparison of signal quality between the investigational device and reference monitor using signal-to-noise ratio analysis. Signal quality is measured in decibels (dB), where higher values indicate cleaner signals with less noise interference. Equivalence is assessed using statistical comparison methods to determine if signal quality differences fall within clinically acceptable ranges.
Device Adhesion Success Rate During Extended Wear | Over 15-day continuous monitoring period
  Percentage of participants who successfully complete the full monitoring period without device adhesion failure. Adhesion failure is defined as device detachment that prevents reliable ECG signal acquisition. Success is measured by the proportion of participants maintaining adequate device adherence throughout the intended wear duration.

CONTACTS AND LOCATIONS:
Locations (1):
- Perin Health Devices, Woodland Hills, California, United States